CLINICAL TRIAL: NCT06475807
Title: Cancer Nutrition Study: CaNS - A Pilot Study of Dietary Interventions in Cancer Patients Treated With Immune Checkpoint Inhibitors
Brief Title: Dietary Interventions in Cancer Patients Treated With Immune Checkpoint Inhibitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Hassane M. Zarour, MD, Professor of Medicine, Immunology, and Dermatology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCC 23-105
Record Dates: First submitted 2024-06-04; First posted 2024-06-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: PD-1/PD-L1 Inhibitors; inflammatory cytokines; gut microbiota
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- high-fermented food + high fiber supplementation (Experimental): Step 1: patients will consume high-fermented food
  Step 2: High fiber supplementation
  Interventions: Dietary Supplement: High-fermented food; Dietary Supplement: High fiber supplementation

INTERVENTIONS:
Dietary Supplement: High-fermented food — Step 1: patients will consume high-fermented food
Dietary Supplement: High fiber supplementation — Step 2: High fiber supplementation

SUMMARY:
This pilot trial will study the potential impact of two distinct dietary interventions with sequential use of high-fermented foods and high-fiber supplements on the gut microbiome and antitumor immunity in patients with melanoma and non-small cell lung cancer (NSCLC) treated with immune checkpoint inhibitors. The trial aims to understand how dietary changes affect the composition and function of the gut microbiome, together with immunological and metabolomic markers in serum in patients with melanoma and NSCLC who are undergoing standard-of-care treatment with a PD-1/PD-L1 Inhibitors (neoadjuvant, adjuvant or consolidation)

DETAILED DESCRIPTION:
Several studies have shown that diet can modulate the gut microbiome and affect the biology of the immune system. The role of the high-fermented food diet and high-fiber supplementation on gut microbiome in patients with cancer treated with immunotherapy will be evaluated. Fermented diet and high-fiber supplementation rational: a high-fermented food diet promotes gut microbiome composition and lowers systemic inflammatory markers. Additionally, high fiber diet may be associated with improved clinical outcomes in immune checkpoint inhibitor treated cancer patients. The effect of high-fermented food and high-fiber supplementation on gut microbiome and systemic inflammation in patients with cancer will be examined. The results of this study will be used to help to design future dietary intervention trials in cancer patients receiving immunotherapy. Baseline diet information, stool and blood samples will be collected. Patients initially receive high-fermented food diet for 4 weeks, followed by 2-week break/observation period and then cross over to high-fiber supplementation for another 4 weeks, followed by 2 weeks break/observation period. During break/observation period patients can eat any type of food, without dietary restrictions. During the dietary intervention period 24-hour dietary recall information will be collected, stool samples weekly and blood sample every 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent.
2. Adult ≥ 18 years of age, willing and able to provide blood and stool specimen and comply with dietary modification, as well as willing to fill out study required questionnaires (paper or electronic and web-based).
3. Patients must have any type of electronic device such as a smartphone, tablet, or computer etc that can access the internet.

   Body mass index (BMI) 18.5-40 kg/m2.
4. Self-reported willingness to adhere with dietary intervention.
5. Self-reported willingness to comply to scheduled follow ups, fill out questionnaires/food logs, provide stool samples and undergo venipuncture
6. Patients who are treated or about to start treatment with standard of care anti-PD-1/PD-L1 therapy will be consented for the dietary intervention study I. Early stage (IIB-IIIC) resected melanoma patient on adjuvant pembrolizumab or nivolumab.

   II. Early stage (IB-IIIA) resected NSCLC patients on adjuvant pembrolizumab or atezolizumab.

   III. Early stage (IB-IIIA) NSCLC patients who are surgical candidates and are treated with neoadjuvant chemotherapy plus immunotherapy (nivolumab or pembrolizumab).

   a. (patients can be enrolled in the study at any point during their treatment period) IV. Stage IIIB or IIIC NSCLC after concurrent chemotherapy and radiotherapy followed by consolidation immunotherapy (durvalumab).

   V. LS-SCLC after concurrent chemotherapy and radiotherapy followed by consolidation immunotherapy (durvalumab)
7. Melanoma patients with stage IIB-IIIC, currently enrolled in a clinical trial and randomized to the standard of care arm (e.g., adjuvant nivolumab or adjuvant pembrolizumab), as permitted by the protocols of the enrolled clinical trial.
8. Melanoma patients with a single metastatic or recurrent lesion who have undergone tumor resection and are currently receiving adjuvant treatment with nivolumab or pembrolizumab.
9. Stage IIB-IIIA NSCLC patients currently enrolled in a clinical trial and randomized to the standard of care anti-PD1/anti-PD-L1 arm after tumor resection or stage IIIB/C NSCLC or LS-SCLC patients after concurrent chemo/RT enrolled in a clinical trial and randomized to the standard of care consolidation immunotherapy arm as permitted by the protocols of the enrolled clinical trial.

Exclusion Criteria:

1. Patients receiving ICIs enrolled in a clinical trial in the experimental arm.
2. Use of any of the following drugs within the last 4 weeks:

   1. Systemic antibiotics, antifungals, antivirals, or antiparasitics (intravenous, intramuscular, or oral);
   2. Oral, intravenous, intramuscular, nasal, or inhaled corticosteroids ((> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study intervention administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease)
   3. Cytokines.
   4. Methotrexate or immunosuppressive cytotoxic agents.
   5. Regularly taking probiotics, fiber supplements, or any other medication or pre-biotic dietary supplement that could affect the study outcome as determined by the principal investigator and unable/unwilling to discontinue for the study. These agents must be discontinued at least 14 days prior to the start of the diet.
3. Current use of chronic alcohol within the last 4 weeks, defined as more than five 1.5-ounce servings of 80-proof distilled spirits, five 12-ounce servings of beer, or five 5-ounce servings of wine per day.
4. Current consumption of fiber >25g (determined based on patient reported intake or baseline DHQ3 assessment) or fermented food ≥≥3 portions a day (foods/drinks tested in the clinical trial, for example coffee beverage is considered to be a fermented drink but will not count towards the consume fermented food intake).
5. Any major bowel resection at any time.
6. Medical contraindications to intervention diet as determined by the treating physician.
7. Systemic antibiotics and proton pump inhibitors (PPis) are not allowable during the study (should be discontinued >21 days prior). If PPIs or systemic antibiotics are initiated by the patient's treating physician, the patient should report this to the study team during the study period.
8. Unable or unwilling to adhere schedule interventions and study procedures.
9. History of active uncontrolled gastrointestinal disorders or diseases, including:

   1. Inflammatory bowel disease (IBD), including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis.
   2. Malabsorption (e.g active celiac disease)
   3. Active Persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent), or Helicobacter pylori infection (untreated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in cell frequency of gut microbiota composition | Up to 14 weeks
  Changes in gut microbiome diversity and function, evaluated with metagenomics, identify differentially abundant taxa and assess all genes in all organisms present in each fecal microbiota sample in pre- vs. post- each dietary using PERMANOVA. This will be measured as change of cell frequency and calculated as percentage change.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | Up to 14 weeks
  Incidence of anti-PD-1/PD-L1 therapy treatment-related grade 3 or more toxicities per CTCAE v5.0
Changes in cell frequency of circulating adaptive immune cells | Up to 14 weeks
  Changes in the circulating adaptive and innate cells in the systemic circulation, evaluated with multiparameter flow cytometry, peripheral blood mononuclear cells will be used to evaluate cell frequency, phenotype, and function. This will be measured as change of cell frequency and calculated as percentage change.

CONTACTS AND LOCATIONS:
Overall Officials: Hassane M Zarour, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No